CLINICAL TRIAL: NCT06116006
Title: fNIRS Study of Effort-dependent Brain Activations During Pointing Movements of the Upper Limb in Post-stroke Patients and Healthy Subjects
Acronym: BIROBONIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique Les Trois Soleils (Other)
Collaborators: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02827-36
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Healthy
Keywords: stroke; upper limb; robot-based therapy; physical modalities; effort; fnirs; cortical activation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with 3 experimental conditions (Other): 3 types of upper limb pointing movements:
  * movements with robot assistance
  * movements without robot assistance
  * movements with robot resistance
  Interventions: Other: Upper limb pointing movements in 3 experimental conditions

INTERVENTIONS:
Other: Upper limb pointing movements in 3 experimental conditions — Recording of cerebral hemodynamic with fNIRS during upper limb pointing movements with a robotic device in three conditions: movements with robot assistance, movements without robot assistance and movements with robot resistance. Each subject are recorded during 6 trials for each condition (18 trials). The order is counterbalanced among the subjects.

SUMMARY:
Background: Following a stroke, as part of neurorehabilitation, the intensity of effort is important to promote neural changes and stimulate motor recovery. There are few studies concerning the cortical activity involved at different levels of intensity during upper limb motor training.

Objective: To investigate cortex activation while walking an exoskeleton with 4 levels of guidance force in healthy controls.

DETAILED DESCRIPTION:
Upper limb paresis is the most common motor deficit following a stroke, and its long-term persistence has an impact on patients' functional recovery and quality of life. Rehabilitation is therefore a major challenge in restoring functional independence.

New physical treatments have been developed over the last 20 years to optimize motor relearning by intensifying motor rehabilitation; among them, therapy using robotic devices has shown its effectiveness in reducing motor deficits.

This therapy offers various options ranging from assistance to movement resistance, which modulates the intensity of effort required of patients during target-pointing exercises.

The brain mechanisms involved in this type of rehabilitation remains imperfectly understood.

Functional neuroimaging techniques such as magnetic resonance imaging (fMRI), positron emission tomography (PET) and functional near-infrared spectroscopy (fNIRS) provide important information on brain activation induced by external stimuli. Among these, fNIRS is a non-invasive method for measuring hemodynamic responses associated with activation of the cerebral cortex. It enables the study of cerebral neurovascular coupling, and is based on the fact that an activated cerebral region increases its oxygen consumption and thus local blood volume and flow.

A better understanding of the cortical effects resulting from the physical forces applied to the upper limb could help optimize the rehabilitation treatment of patients, thereby promoting cerebral plasticity.The aim of the study is to compare cortical responses measured by fNIRS during 3 types of upper limb pointing movement:

* robot-assisted movements
* robot-unassisted movements
* robot-resisted movements

in patients with chronic hemiparesis after stroke and in healthy subjects.

ELIGIBILITY:
INCLUSION CRITERIA

For stroke subjects

* Age ≥18 years;
* Stroke-induced hemiparesis, chronic phase (>6 months post-stroke);
* Moderate upper limb paresis defined by an upper limb FMA score 20 pts < FMA score < 47 pts ;
* Right-handed patient;
* Patient having agreed to sign an informed consent form;
* Patient affiliated to the French social security system.

For healthy subjects

* Age-matched participant, for each stroke subject included will be associated a control subject of the same age (to the nearest 5 years);
* Right-handed participant;
* Participant having agreed to sign an informed consent form;
* Participant affiliated to the French social security system.

NON-INCLUSION CRITERIA

For stroke subjects

* Cognitive impairment making participation in the study impossible;
* Phasic disorders preventing comprehension of instructions and effective communication.

For healthy subjects

* Pathology of the dominant upper limb;
* Cognitive disorders making participation in the study impossible;
* Presence of labelled or unlabelled neurological disorders;
* Persons under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of oxyhemoglobin concentration during upper limb tasks | Day 0
Change of desoxyhemoglobin concentration during upper limb tasks | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- La Clinique Les Trois Soleils, Boissise-le-Roi, France

REFERENCES:
- [Background] Shi P, Li A, Yu H. Response of the Cerebral Cortex to Resistance and Non-resistance Exercise Under Different Trajectories: A Functional Near-Infrared Spectroscopy Study. Front Neurosci. 2021 Oct 13;15:685920. doi: 10.3389/fnins.2021.685920. eCollection 2021. PMID 34720845
- [Background] Zheng J, Shi P, Fan M, Liang S, Li S, Yu H. Effects of passive and active training modes of upper-limb rehabilitation robot on cortical activation: a functional near-infrared spectroscopy study. Neuroreport. 2021 Apr 7;32(6):479-488. doi: 10.1097/WNR.0000000000001615. PMID 33788815